CLINICAL TRIAL: NCT03861195
Title: Comparative Prospective Data Collection in Connection With Two Different Treatment Methods: Robotic Assisted Laparoscopy and Conventional Laparoscopy
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: MT_SOS I
Record Dates: First submitted 2019-02-21; First posted 2019-03-04 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-02

CONDITIONS: Uterine Diseases
MeSH Terms: conditions — Uterine Diseases | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Da Vinci Robotic Surgical System
  Interventions: Procedure: laparoscopic surgery
- conventional laparoscopic surgery
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: laparoscopic surgery — patients affected by uterine diseases that undergo treatment

SUMMARY:
This is a prospective, randomized, single-center, observational clinical trial at the Department of Women's Health of the University Clinic Tübingen. Four hundred patients affected by uterine diseases that undergo treatment with robotic assisted laparoscopic procedures using the Da Vinci Robotic Surgical System (200 patients) or conventional laparoscopic surgery (200 patients) will be recruited. In addition retrospective data of 200 patients that underwent conventional laparoscopic surgery in the past will be documented. At the end of patient recruitment, surgical procedure times, the technical limits encountered, estimated blood loss, intra- and post-operative complications and the percentage of conversions from the robotic assisted treatment /conventional laparoscopic surgery to multiple access and/or to a laparotomic (open) approach will be documented.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* BMI ≤40 kg/m2
* indication for hysterectomy for benign disease or prophylactic surgery due to hereditary cancer
* indication for radical hysterectomy and/or pelvic-/para-aortic (sentinel-node) lymphadenectomy for cervical cancer
* indication for modified radical hysterectomy and/or pelvic-/para-aortic (sentinel-node) lymphadenectomy for endometrial cancer
* size of uterus and vagina allows for retrieval by the vaginal route in cancer patients
* written informed consent

Exclusion Criteria:

* known extensive intra-abdominal adhesions
* anaesthesiological contraindications to laparoscopy
* women with pacemaker or other implants where electrosurgery is to be avoided
* women with known defects of the hemostasis
* pregnancy
* other internal or anatomical criteria that preclude a minimal invasive approach
* inability to understand patient information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
operative time | 60 minutes
  (minutes from first incision to skin closure)
time under narcosis | 60 minutes
console time | 60 minutes
estimated blood loss (milliliters) | 60 minutes
  using the following formula: ((Hemoglobin concentration preoperative (g/l)) - (Hemoglobin 1st day postoperative (g/l)))/((Hemoglobin preoperative (g/l)) - (Hemoglobin 1st day postoperative (g/l)))/2) × 1000
conversion to other surgical procedures | 60 minutes
time to discharge | 60 minutes
intraoperative complications | 60 minutes
  occurring during the surgical procedure
perioperative complications | 24 hours
  occurring less than 24h after the surgical procedure, according to the Clavien-Dindo classification of surgical complications
postoperative complications | 6 months
  occurring more than 24h after the surgical procedure up to 6 months after surgical procedure, according to the Clavien-Dindo classification of surgical complications
German version of the Short Form-36health survey questionnaire Medical Outcomes Trust | 3 and 6 months
  Medical Outcomes Trust: SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting.
German version of the female sexual function index (FSFI) questionnaire | 3 and 6 months
  female sexual function index: a multidimensional self-report instrument for the assessment of female sexual function

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tuebingen, Department of Women's Health, Tübingen, Germany